CLINICAL TRIAL: NCT07286175
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Parallel-Arm Study to Investigate the Efficacy and Safety of Adjunctive Treatment With Brenipatide in Delaying Time to Relapse Compared With Placebo in Adult Participants With Bipolar Disorder (RENEW-Bipolar-1)
Brief Title: A Study of Brenipatide in Adult Participants With Bipolar Disorder (RENEW-Bipolar-1)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27365; J2S-MC-GZMJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-11-21; First posted 2025-12-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brenipatide Dose 1 (Experimental): Brenipatide administered subcutaneous (SC) + SoC.
  Interventions: Drug: Brenipatide
- Brenipatide Dose 2 . (Experimental): Brenipatide administered subcutaneous (SC) + SoC.
  Interventions: Drug: Brenipatide
- Placebo (Placebo Comparator): Placebo administered SC + SoC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brenipatide — Administered SC
  Other Names: LY3537031
  Arms: Brenipatide Dose 1; Brenipatide Dose 2 .
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of brenipatide when administered with standard of care (SoC), compared with placebo plus SoC in delaying the worsening of bipolar disorder symptoms.

The trial is divided into three periods as follows: Screening period that will last approximately 1 month, treatment period that will last a minimum of 6 months, and the follow up period that will last approximately 2 months. The duration of study participation may vary and may be shortened if bipolar symptoms worsen or if withdrawal from the study occurs for any reason.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for bipolar disorder I or bipolar disorder II
* Are reliable and willing to make themselves available for the duration of the study and attend required study visits, and are willing and able to follow study procedures as required, such as

  * self-inject study intervention
  * store and use the provided blinded study intervention, as directed
  * maintain electronic and paper study diaries, as applicable, and
  * complete the required questionnaires
* Are on stable standard of care medication for bipolar disorder

Exclusion Criteria:

* Have a lifetime history or current diagnosis of the following according to DSM-5 criteria:

  * schizophrenia or other psychotic disorder
  * borderline personality disorder, or
  * any eating disorder
* Have type 1 diabetes mellitus, or a history of

  * ketoacidosis, or
  * hyperosmolar state or coma
* Have evidence of moderate or severe substance or alcohol use disorder within the past 180 days prior to screening
* Are actively suicidal and or deemed to be at significant risk for suicide
* Have participated in a clinical study and received active treatment, or unknown if they received active treatment, within 90 days or 5 half-lives (whichever is longer) before screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Time to Relapse Defined as Days from Randomization to the Date on Which the Participant Meets Any Relapse Criterion | Randomization up to at least 6 months

SECONDARY OUTCOMES:
Change from Baseline in Sheehan Disability Scale (SDS) Global Functional Impairment Score | Baseline, up to at least 6 months
Change from Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score | Baseline, up to at least 6 months
Change from Baseline in Young Mania Rating Scale (YMRS) Total Score | Baseline, up to at least 6 months
Change from Baseline in Recovering Quality of Life - 20 Items (ReQoL-20) Total Score | Baseline, up to at least 6 months
Change from Baseline in Patient Rated Outcome as Measured by Patient's Global Impression of Severity (PGI-S) | Baseline, up to at least 6 months
Mean Percent Change in Body Weight in Participants with a Baseline Body Mass Index (BMI) of ≥25 kg/m2 | Baseline, up to at least 6 months
Mean Percent Change in Body Weight in Participants with a Baseline Body Mass Index (BMI) of ≥25 kg/m2 and on an Atypical Antipsychotic | Baseline, up to at least 6 months
Pharmacokinetic (PK): Average Steady State Plasma Concentration (Cavg) of Brenipatide | Baseline, up to at least 6 months
Number of Participants with Treatment-Emergent Anti-Drug Antibodies | Baseline, up to at least 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (85):
- United States (20):
  - ATP Clinical Research, Orange, California
  - Yale University School of Medicine, New Haven, Connecticut
  - AGA Clinical Trials, Hialeah, Florida
  - Accel Research Sites - Maitland Clinical Research Unit, Maitland, Florida
  - K2 Medical Research - Maitland, Maitland, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - CLA Research, Naples, Florida
  - Charter Research - Orlando, Orlando, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Covenant Medical Center, Waterloo, Iowa
  - CBH Health, Gaithersburg, Maryland
  - Elixia MA, Springfield, Massachusetts
  - Adams Clinical Watertown, Watertown, Massachusetts
  - Penn Medicine: University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Revival Research Institute, LLC, McKinney, Texas
  - Pillar Clinical Research - Richardson, Richardson, Texas
  - Alpine Research Organization, Clinton, Utah
  - Re:Cognition Health, Fairfax, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Argentina (12):
  - Hospital Italiano de Buenos Aires, ABB
  - Centro Neurobiológico y de Estrés Traumático (CENydET), Buenos Aires
  - Instituto Nacional de Psicopatología (INAPsi)- FunDaMos, Buenos Aires
  - Stat Research S.A., Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - Instituto Médico DAMIC, Córdoba
  - Instituto Kremer, Córdoba
  - Centro Médico Luquez, Córdoba
  - Global Psy Asociación Civil, La Plata
  - Fundacion Scherbovsky, Mendoza
  - INECO Neurociencias Oroño, Rosario
  - Clinica El Jardin, Santiago del Estero
- Brazil (9):
  - Chronos Pesquisa Clínica, Brasília
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - Centro de Pesquisa Clínica de Marília - CPCLIM, Marília
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Facili Centro Integrado de Psiquiatria, São Bernardo do Campo
  - CPQuali Pesquisa Clínica, São Paulo
  - BR Trials - Ensaios Clinicos e Consultoria, São Paulo
  - Clinica Viver - Centro de Desospitalizacao Humana, São Paulo
  - A2Z Clinical Centro Avançado De Pesquisa Clínica - Valinhos, Valinhos
- China (10):
  - The Second People's Hospital of Hunan Province, Changsha
  - The Seventh People's Hospital of Hangzhou, Hangzhou
  - 3rd People's Hospital of Huzhou, Huzhou
  - Shangdong Mental Health Center, Jinan
  - Shanghai Mental Health Center, Shanghai
  - Shanghai Tongji Hospital, Shanghai
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Anding Hospital, Tianjin
  - Xiamen Xianyue Hospital, Xiamen
  - Zhumadian Psychiatric Hospital, Zhumadian
- India (10):
  - Galaxy Superspeciality Hospital, Aurangabad
  - Belagavi Institute of Medical Sciences - Belagavi, Belgavi
  - All India Institute of Medical Sciences (AIIMS) - Bhopal, Bhopal
  - Society for Psychiatric Update and Research, Chhatrapati Sambhajinagar
  - Dr. Ram Manohar Lohia Institute of Medical Sciences, Lucknow
  - Career Institute of Medical Sciences and Hospital - Lucknow, Lucknow
  - Assured Care Plus Hospital, Nashik
  - Lifepoint Multispeciality Hospital, Pune
  - Sowmanasya Hospital and Institute of Psychiatry, Tiruchirappalli
  - Deva Institute Of Healthcare Research, Varanasi
- Japan (15):
  - Uematsu Mental Clinic, Chikugo
  - Jimbocho Mental Clinic, Chiyoda City
  - Horikoshi Mental Somatic Clinic, Fukushima
  - Saitama Medical University Hospital, Iruma
  - Rainbow and Sea Hospital, Karatsu
  - Monzen-nakacho Mental Clinic, Kōtō City
  - Suizenji Life Clinic, Kumamoto
  - Kure Medical Center, Kure
  - Hirota Clinic, Kurume
  - Yutaka Clinic, Sagamihara
  - Maynds Tower Mental Clinic, Shibuya-ku
  - Himorogi Psychiatric Institute - Tokyo - Ichigayatamachi, Tokyo
  - Ikebukuro Olive Mental Clinic, Toshima City
  - Yamagata Sakuracho Hospital, Yamagata
  - Miki Mental Clinic, Yokohama
- Mexico (8):
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara
  - B&B Investigaciones Medicas S.C., Mazatlán
  - Centro de Investigación Clinica Chapultepec, Mexico City
  - Ketamine Clinic México, Mexico City
  - Medical Care and Research SA de CV, Mérida
  - Centro de Investigacion Clinica Chapultepec, Morelia
  - Instituto Jalisciense de Salud Mental, Zapopan
- SCB Research Center, Bayamón, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Brenipatide in Adult Participants With Bipolar Disorder (RENEW-Bipolar-1) — https://trials.lilly.com/en-US/trial/674575